CLINICAL TRIAL: NCT01972204
Title: A Study About the Impact of Intensive Instruction on the Use of Aricept and the Reasons for Discontinuation in Patients With Alzheimer's Disease
Brief Title: Intensive Instruction on the Use of Aricept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mirai Iryo Research Center, Inc. (Other)
Responsible Party: Principal Investigator, Tetsumasa Kamei, Hospital Director, Mirai Iryo Research Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART-2013-01
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Alzheimer's Type Dementia

ARMS (2):
- Intensive adherence instruction (Experimental): Intensive adherence instruction group will receive 5 visits and receive the instruction on the use of Aricept with educational brochure
  Interventions: Behavioral: Intensive adherence instruction
- Control (Sham Comparator): The control group will receive 5 visits and receive the instruction on the use of Aricept as per usual practice.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intensive adherence instruction — Instruction with educational brochure
  Arms: Intensive adherence instruction
Behavioral: Control — Instruction as per usual practice
  Arms: Control

SUMMARY:
The purpose of this study is to examine the influence of the instruction on the use of Aricept with educational brochure on the 48-week medication persistence and to assess the reasons for discontinuation.

DETAILED DESCRIPTION:
To examine the influence of the instruction on the use of Aricept with educational brochure comparing to the ordinary instruction on the 48-week medication persistence and to assess the reasons for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic evidence of probable Alzheimer's type Dementia consistent with DSM-IV.
* Written informed consent will be obtained from subject (if possible) or from the subject's legal guardian or other representative (according to Japanese regulations as appropriate) prior to beginning screening activities.
* Patients having caregivers who submit written consent for cooperative involvement in this study, can provide patients' information necessary for this study, assist treatment compliance, and escort patients on required visits to study institution.
* Outpatients in their own home.

Exclusion Criteria:

* Patients treated with donepezil, galantamine, rivastigmine in 4 weeks immediately before enrollment.
* Known hypersensitivity to donepezil or piperidine derivatives.
* Involvement in any other investigational drug clinical trail during the preceding 12 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-09; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tetsumasa Kamei, Principal Investigator — Shonan Fujisawa Tokushukai Hospital
Locations (1):
- Shonan Fujisawa Tokushukai Hospital, Fujisawa, Kanagawa, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive Adherence Instruction | Control
Started | 62 | 63
Completed | 58 | 59
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Adherence Instruction | Control | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 58 | 58 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.7 (7.23) | 80.2 (6.99) | 79.9 (7.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 31 | 68
  Male | 21 | 28 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 58 | 59 | 117
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 58 | 59 | 117
Treatmnent for alzheimer's disease before study [Number; unit: participants] | 44 | 48 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Medication Continuation
Description: Number of Participants who Continue the Medication for 48 weeks
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Intensive Adherence Instruction | Control
Number analyzed (Participants) | 58 | 59
participants | 36 | 39

2. Secondary Outcome: Reasons for Discontinuation
Description: Reasons for discontinuation of the Medication
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Adherence Instruction | Control
Number analyzed (Participants) | 22 | 20
Participants
  Pysician's decision | 17 | 11
  Participant's wish | 2 | 4
  Caretaker's wish | 3 | 5

3. Secondary Outcome: Number of Participants With Medication Discontinuation Due to Change to Alicept or Generics
Description: Number of Participants who descontinue the Clinical Trial Medication due to Change to Alicept (not for clinical trial) or Generics
Time Frame: 48 weeks
Measure: Number; unit: participants
Arm/Group | Intensive Adherence Instruction | Control
Number analyzed (Participants) | 58 | 59
participants | 5 | 7

4. Secondary Outcome: Adverse Events
Description: Adverse Events for each arm
Time Frame: Week 2, 12, 24, 48
Measure: Number; unit: participants
Arm/Group | Intensive Adherence Instruction | Control
Number analyzed (Participants) | 58 | 59
participants | 33 | 23

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intensive Adherence Instruction | Control
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/59
Other Adverse Events (participants affected / at risk) | 20/58 | 14/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Adherence Instruction (N=58) | Control (N=59)
nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5)
contusion (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
hypertention (Vascular disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT01972204/Prot_SAP_000.pdf